CLINICAL TRIAL: NCT02291900
Title: Talar Avascular Necrosis: Surgical Angiogenesis Compared to Core Decompression With Osseous Auto Grafting
Brief Title: Talar Avascular Necrosis: Surgical Angiogenesis vs. Core Decompression
Acronym: TalarAVN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: BG Trauma Center Ludwigshafen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BGU - 01/14
Record Dates: First submitted 2014-11-12; First posted 2014-11-17 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Avascular Necrosis of Bone
Keywords: avascular necrosis, talus, medial femoral condyle
MeSH Terms: conditions — Osteonecrosis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- medial femoral condyle (Active Comparator): Patients in this arm receive core decompression followed by free vascularized medial femoral condyle graft
  Interventions: Procedure: core decompression
- core decompression (Active Comparator): Patients in this arm receive core decompression followed by osseous autograft from the iliac crest
  Interventions: Procedure: core decompression

INTERVENTIONS:
Procedure: core decompression — retrograd drilling of the avascular talar necrosis, followed by osseous autograft

SUMMARY:
The purpose of this study is to determine if surgical angiogenesis performed in talar avascular necrosis by free microvascular bone grafts from the femoral condyle is a superior technique compared to core decompression and nonvascularized osseous autografts.

DETAILED DESCRIPTION:
The aim of this prospective randomized clinical trial is the comparison of two surgical treatment options for talar avascular necrosis (analogical to Ficat and Arlet stage II and III). The randomized study design allows direct comparability of the outcome after either core decompression and nonvascularized osseous autografting from the iliac crest or core decompression and osseous autografting with a free microvascular medial femoral condyle.

Talar avascular necrosis is caused by osseous malperfusion leading to malnutrition and destruction of the talar bone. The extend of this malperfusion is variable and can be categorized in 4 stages. The osseous defects can remain without consequences (stage I) or lead to irreversible talar destruction. The current treatment option for stage II and III is the core decompression followed by osseous auto grafting from the iliac crest. Reducing the intraosseal pressure and filling the drill holes with the bone graft can lead to reperfusion of the talus.

A new technique is to fill the drill hole with a vascularized bone graft from the medial femoral condyle, using microvascular anastomosis. This procedure has already been approved for the treatment of avascular necrosis and malperfusion of the carpus (lunate and scaphoid) as well as the femoral head.

Patients are examined preoperative as well as 3, 6 and 12 month after operation, documenting the active range of motion and pain sensation while resting and on activity. Well established scores like the AOFAS Ankle-Hindfoot Score and the Lower Extremity Functional Scale are used to get subjective and objective informations about patients' daily life and postoperative satisfaction. X-Rays are taken at the same stages. MRIs of the ankle joint with contrast agent are performed before as well as 6 and 12 months after surgery.

Statistical analysis is performed using the Statistical Package for the Social Sciences (SPSS). The Study protocol has been approved by the Ethics Commission of Rheinland-Pfalz. Interventions are done according to the declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* Avascular talar necrosis stage 2 and 3 (Ficat and Arlet)
* signed patient consent form

Exclusion Criteria:

* steroid or chemo therapy
* participation in a different study
* pregnancy
* peripheral artery occlusive disease stage 3 and 4
* avascular talar necrosis stage 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-02; Primary Completion 2015-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Pain reduction | 3, 6, 12 months post operation

SECONDARY OUTCOMES:
Lower Extremity Functional Scale | pre operation; 3, 6, 12 month post operation
Revascularization (Association International de Recherche sur la Circulation Osseuse-Criteria) | 6 and 12 month postoperative
American Orthopaedic Foot and Ankle Society- Ankle and Hindfoot Score | pre operation; 3, 6, 12 month post operation

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Kneser, Phd, MD, Study Chair — BG Trauma Center Ludwigshafen
Locations (1):
- BG Trauma Center Ludwigshafen, Ludwigshafen am Rhein, Rhineland-Palatinate, Germany